CLINICAL TRIAL: NCT06504264
Title: The Effect of Articulatory Gestures on Word Reading, Non-word Reading, and Phonemic Segmentation in 4-year Olds
Brief Title: The Effect of Articulatory Gestures on Early Literacy Skills in 4-year Olds
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montclair State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB-FY23-24-3843
Record Dates: First submitted 2024-07-03; First posted 2024-07-16 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Early Literacy; Articulatory Gestures; Phonemic Awareness
MeSH Terms: conditions — Literacy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LPA: Letters-phonemes-articulatory gestures (Experimental): This group will receive training for phonemic segmentation that includes using printed letters, sounds (phonemes) while simultaneously learning the articulation placements of the letters/sounds.
  Interventions: Behavioral: phonemic segmentation
- LPM: Letters-phonemes-general mouth awareness (Experimental): This group will receive training for phonemic segmentation that includes using printed letters, sounds (phonemes) while simultaneously learning about the mouth in general.
  Interventions: Behavioral: phonemic segmentation
- LP: Letters-phonemes (Experimental): This group will receive training for phonemic segmentation that includes using printed letters and sounds (phonemes) only.
  Interventions: Behavioral: phonemic segmentation

INTERVENTIONS:
Behavioral: phonemic segmentation — during phonemic segmentation activities, articulatory gestures will be used while teaching letters and their sounds.

SUMMARY:
This study will use an experimental design to explore if articulatory gestures (with letters and phonemic awareness training) enhance early literacy skills more than general mouth awareness training (with letters and phonemic awareness training) or letter/phonemic awareness training alone.

DETAILED DESCRIPTION:
Multisensory reading strategies, which recruit one or more of the five senses, are routinely used in general education classrooms as well as with children who are struggling readers. Despite their wide use in schools, little research exists to substantiate the utilizing these strategies to enhance literacy. One type of multisensory reading strategy, articulatory gestures, is of particular interest to speech-language pathologists (SLPs) as they are uniquely positioned to provide speech sound placement cues. Limitations of the few prior studies that exist have prevented the isolation of the articulatory gestures themselves as the main contributor to the gains seen in literacy. This study aims to control for factors such as motivation, engagement, and time on task to explore the specific contribution of articulation strategies during phonemic awareness training on phoneme segmentation, reading of phonemically spelled words, and nonword reading in typically developing four-year old children. Using an experimental design, participants will be randomly assigned to one of three conditions: 1) phonemic awareness training with articulatory gestures, 2) phonemic awareness training with general mouth pictures, and 3) phonemic awareness training with no mouth/articulation pictures at all. Interventions will focus on phoneme-letter correspondence and phonemic segmentation using strategies specific to each group and differences between groups will be considered for pre and posttest measures.

ELIGIBILITY:
Inclusion Criteria:

* Knows 15 letter names
* Passes hearing screening
* Passes Fluharty-2 Language Screening
* Can segment no more than three consonant-vowel (CV), VC, or CVC words into phonemes
* Not able to read more than one word or nonword used in the posttest.

Exclusion Criteria:

* Does not know 15 letter names
* Fails hearing screening
* Fails Fluharty-2 Language Screening
* Can segment more than three consonant-vowel (CV), VC, or CVC words into phonemes
* Reads more than one word or nonword used in the posttest.

Ages: 48 Months to 59 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 9 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
number of words correctly phonemically segmented from primary investigator created list | immediately after the intervention
  will tell the sounds in 9 words presented orally

SECONDARY OUTCOMES:
number of words read correctly from primary investigator created list | immediately after the intervention
  will read phonemically 6 spelled words
number of nonwords read correctly from primary investigator created list | immediately after the intervention
  will read 7 nonwords

CONTACTS AND LOCATIONS:
Overall Officials: Robyn Becker, Principal Investigator — Montclair State University
Locations (1):
- Montclair State University, Montclair, New Jersey, United States

IPD SHARING:
Plan to Share IPD: No